CLINICAL TRIAL: NCT06289712
Title: Evaluation of the Ablation of Hepatic Lesions by Electroporation
Acronym: EVALHEP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Inria Team MONC (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP231660
Record Dates: First submitted 2024-02-23; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Liver Cancer
Keywords: Liver cancer; Hepatocellular Carcinoma; Irreversible Electroporation
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Irreversible electroporation is a curative treatment for cancerous liver lesions, performed on deep-seated tumors that are not eligible for surgical resection or percutaneous thermal ablation.

The EVALHEP project aims to develop criteria for evaluating the effectiveness of the treatment based on imaging, mathematical models, and numerical simulations to assist radiologists who perform these complex procedures.

DETAILED DESCRIPTION:
Percutaneous destruction of malignant liver tumors has been developing in routine clinical practice for around twenty years, and is performed by interventional radiologists under imaging guidance (ultrasound, computed tomography (CT), Cone-Beam CT...).

Irreversible electroporation (IRE) is a percutaneous tumor destruction technique distinguished from other ablation methods by its non-thermal mechanism of action. The rationale behind IRE is that cells subjected to a powerful pulsed electric field will have their membrane irreversibly damaged and destroyed, while the surrounding extracellular matrix will be respected. This technology offers the opportunity to effectively destroy lesions that would be impossible to treat by any other method, due to their critical tumor location, close to vital structures at risk.

Although it has demonstrated its clinical efficacy over the years, with the potential to provide safe, curative treatment for patients with deep, poorly located tumors, IRE is considered a complex procedure, subject to numerous variability factors, and remains under-utilized to this day. Precise insertion of several needles (up to 6) at tumor level is required to obtain a homogeneous electric field of sufficient intensity. To date, there is no way of assessing the effectiveness of the procedure in real time, and inaccuracies in needle positioning or in treatment parameters will generate changes in the distribution of the electric field that may adversely affect treatment efficacy. What's more, it remains difficult to assess treatment efficacy on post-therapy images, the interpretation of which is subject to controversy.

The Interventional Radiology (IR) unit of the University Hospitals of Paris Seine Saint Denis (HUPSSD) has been using IRE for over 10 years as part of its clinical routine, mainly for the ablation of liver tumors, and in particular hepatocellular carcinoma (HCC) which is inoperable and ineligible for conventional thermo-ablation. Over the past ten years, more than 350 patients have benefited from one or more IREs for the treatment of liver tumors at HUPSSD, making the department a reference center in the field.

Thanks to the contributions of mathematics applied to oncology, numerical tools and the clinical experience of the HUPSSD IR department, the aim of this project is to develop evaluation criteria for IRE ablations of liver tumors based on clinical imaging and numerical simulations of the electric field.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Informed patients who have not objected to participating in the research, or in the case of deceased patients, who have not objected to the processing of their data during their lifetime.
* Diagnosis of malignant liver tumor based on either :

  * Anatomopathological analysis based on an image-guided biopsy prior to surgery (or performed during surgery and contributing to the diagnosis).
  * Criteria for non-invasive diagnosis of HCC on pre-procedural imaging: CT and/or MRI with contrast injection demonstrating tumor enhancement kinetics after injection typical of HCC (arterial contrast and portal and/or late lavage of a tumor over 10 mm in the presence of chronic liver disease, EASL criteria) and/or Li-RADS 5 classification.
* Percutaneous removal of liver tumor by Irreversible Electroporation (IRE) performed during the study period.
* Complete peri-interventional imaging file including:

  * CT and/or MRI of the liver with contrast injection performed within 3 months prior to the procedure
  * Early liver MRI within 4 days of procedure
  * Post-treatment hepatic MRI performed 3 to 6 weeks after the IRE procedure
* Cone-Beam CT (CBCT) volume reconstructions acquired during the IRE procedure available and including at least :

  * An initial acquisition before electrode placement
  * An acquisition with the electrodes in place in their final position
* Per-procedural data recorded in the available IRE generator, including the number of electrodes, their schematic spatial configuration, pulse data with test pulses, applied potential (Volt) and measured currents (Amperes) between each electrode combination.

Exclusion Criteria:

* Contraindications to MRI:

  * Implantable cardiac pacemaker or defibrillator not compatible with MRI, neurostimulator, cochlear implant, intra-cerebral ferromagnetic vascular clips, intraocular or cerebral metallic foreign bodies, insulin pump
* Contraindication to percutaneous IRE treatment due to :

  * the presence of uncontrolled cardiac rhythm disorders
  * Presence of a Pacemaker or implantable cardioverter defibrillator
* Absence of CBCT volume images of the IRE needles in their final position (or modification of their position between the time of CBCT acquisition and delivery of the electrical impulses).
* If the tumor treated corresponds to a remnant after another locoregional treatment modality (but inclusion possible if the tumor treated corresponds to a local recurrence if it was discovered more than 4 months after a locoregional treatment deemed complete).
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cancer (hepatocellular carcinoma) treated by IRE between 2022 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
Correlate 3D numerical simulations of the IRE electric field with patient imaging follow-up | 72 hours and 1 month after treatment
  Demonstrate a correlation between the treatment zones segmented on post-therapy MRI scans and the three-dimensional electric field isolines obtained using digital simulations.

SECONDARY OUTCOMES:
Calculation of the tumor coverage rate by the various electric field isolines at different relevant values (for example, three-dimensional isolines between 300 and 700V.cm-1 will be simulated numerically). | 72 hours and 1 month after treatment
  Determine a threshold for IRE of liver tumors by combining numerical electric field resolution and post-treatment imaging data.
Correlation of recovery rate with treatment outcome and local recurrence during clinical follow-up | 72 hours and 1 month after treatment
  Assess inter-individual variations in liver and tumor conductivity values based on impedance data provided by the IRE generator.
Identification and assessment of imaging biomarkers (radiomics-based) using numerical simulation and post-therapeutic imaging for treatment response evaluation. | 72 hours and 1 month after treatment
  Determine a threshold electric field value to be reached for complete treatment (calculation of sensitivity, specificity, PPV, NPV, ROC curve)
Digital resolution of electrical potential and tissue conductivity values from test pulses at the start of the procedure. | 72 hours and 1 month after treatment
  Evaluate the most suitable and clinically relevant numerical electroporation model (linear/non-linear, static/dynamic).
Develop software solutions potentially usable in real-time and tailored for clinical use. | 72 hours and 1 month after treatment
  Demonstrate a correlation between the treatment zones segmented on post-therapy MRI

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SUTTER, Pr,MD, PhD, Study Director — Assistance Publique de Paris
Locations (1):
- Service d'imagerie diagnostique et interventionnelle tri-site des HUPSSD, Bobigny, France

IPD SHARING:
Plan to Share IPD: No